CLINICAL TRIAL: NCT06357221
Title: A Multi-center, Open-label, In-use Study to Assess Efficacy and Tolerability of Topical Skincare Products on Psoriasis Patients
Brief Title: A Study to Assess Efficacy and Tolerability of Topical Skincare Products on Psoriasis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.035
Record Dates: First submitted 2024-03-20; First posted 2024-04-10 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Plaque Psoriasis; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — cetyl alcohol, propylene glycol, sodium lauryl sulfate non-lipid cleansing lotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Skincare Product Treatment (Experimental): Subjects will use topical skincare products to assigned side of the body, per randomization.
  Interventions: Drug: Cetaphil

INTERVENTIONS:
Drug: Cetaphil — Subjects will clean the skin with Cetaphil Gentle Skin Cleanser, and apply Cetaphil Moisturizing Cream to the lesion areas at least twice daily. Subjects will use Cetaphil Daily Facial Moisturizer SPF 35 as needed.
  Other Names: Topical Skincare Treatment

SUMMARY:
Subjects having mild-to-severe plaque psoriasis, with active target lesion plaques, and currently on or starting a prescription treatment for plaque psoriasis will apply a topical skincare regimen to one side of the body. Evaluations of the regimen's efficacy will be conducted at 2 weeks, 4 weeks, and 8 weeks post-baseline.

DETAILED DESCRIPTION:
This is a multi-center, open-label, in-use study. Adult subjects having mild-to-severe plaque psoriasis, with active target lesion plaques, and currently on or starting a prescription treatment for plaque psoriasis will be recruited for participation in the study.

Subjects will report to the site at Baseline (day 0) visit, will be given an informed consent form, HIPAA form, photography release form, and medical history form to complete.

Subjects will be screened on the basis of the selection criteria for study qualification. Eligible subjects will be assessed at Baseline visit and instructed to start applying the skincare products to the assigned side of the body based on the pre-determined randomization.

Subjects to return to the site at Week 2 (± 3 days), Week 4 (± 5 days), and Week 8 (± 5 days) for follow-ups.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 18 years and above
2. Females or males
3. Any Fitzpatrick skin types I-VI, with effort to include n = 2 for each category
4. Any races, with effort to include minimum 10% minority (n = 4) such as American Indian or Alaska Native, Eastern/Southeastern Asian, South Asians, Black or African American, Native Hawaiian or Other Pacific Islander.
5. Any ethnicities, with effort to include minimum 10% (n = 4) of Hispanic, Latino, or Spanish origin
6. Having active target lesion plaques, with minimum area of 2 cm x 2 cm
7. Having mild-to-severe plaque psoriasis with at least 3% Body Surface Area (BSA) and cumulative Target Lesion Severity Score (TLSS) ≥ 6.
8. Currently on or starting a plaque psoriasis prescription treatment such as biologics, oral or topical therapy for psoriasis, or UV therapy.
9. Subject in general good health
10. Subject willing to stop using current topical skincare products during the duration of the study.
11. Subject willing to replace current skincare products with study products for the duration of the study.
12. For female subjects of childbearing potential, she must not be pregnant, breastfeeding or planning pregnancy during the course of the study. Subjects must be willing to take a urine pregnancy test (UPT) at Baseline visit. (Females of non-childbearing potential, e.g., post-menopausal (absence of menstrual bleeding for 1 year without any other medical reason), hysterectomy, or bilateral ovariectomy, are not required to have a UPT.)
13. Ability of giving consent for participation in the study
14. Willing to sign a photography release, with minimum 80% of total study panel
15. Agreement to adhere to the procedures and requirements of the study and to report to the site on the day(s) and at the time(s) scheduled for the assessments

Exclusion Criteria:

1. Pregnant, breastfeeding, or planning pregnancy during the course of the study.
2. Subjects with any known allergies or hypersensitivity to any cosmetics, personal care products, and/or fragrances.
3. History of cancer within the past 5 years
4. History or presence of any skin condition/disease, besides plaque psoriasis, that might interfere with the diagnosis or evaluation of study parameters at the discretion of the investigator.
5. Planning on having surgeries and/or invasive medical procedures during the course of the study
6. Treatment with chemotherapy, immunosuppressive agents, prescription corticosteroids for psoriasis, immunomodulatory therapy (e.g., monoclonal antibodies or antiviral treatment for human immunodeficiency virus or hepatitis C)
7. History or presence of any medical condition that, in the opinion of the Investigator, would make the subject unsuitable for inclusion (e.g., a chronic, relapsing, or hereditary disease that may interfere the outcome of the study).
8. Other condition preventing the subject from entering the study in the Investigator's opinion, (e.g., subjects failing baseline assessments, subjects not likely to avoid other treatments in the treated areas, subjects anticipated to be unavailable or incapable of understanding the study assessments or having unrealistic expectations of the treatment result).
9. Study site personnel, close relatives of the study site personnel (e.g., parents, children, siblings, or spouse), or employees and close relatives of employees at the Sponsor company.
10. Participation in any interventional clinical study within 30 days of screening or planning to participate in another interventional clinical research study while enrolled in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Change in psoriatic Body Surface Area compared to baseline | Baseline, Week 2, Week 4, Week 8
  Body Surface Area is a measure of how much skin is impacted by psoriasis using the following measurement.7 One handprint is equal approximately to 1% of Body Surface Area. A decrease in scores indicates an improvement.
Change in target lesion severity compared to baseline | Baseline, Week 2, Week 4, Week 8
  Target lesion severity will be measured by the Target Lesion Severity Score. Target Lesion Severity Score assesses erythema, induration, and scaling separately on a scale of 0-8, with 0 meaning no evidence of the parameter and 8 meaning very severe presence of the parameter. Target Lesion Severity Score is calculated as cumulative total of all 3 parameters, which a maximum score of 24 (8 x 3). A decrease in scores indicates an improvement.
Change of Physician Global Assessment compared to baseline | Baseline, Week 2, Week 4, Week 8
  Physician Global Assessment assesses overall severity of psoriasis on a scale of 0 to 5, with 0 meaning no presence of psoriasis and 5 meaning very severe presence of psoriasis. A decrease in scores indicates an improvement.
Change in skin quality measured by macroscopic imaging | Baseline, Week 2, Week 4, Week 8
  Macroscopic imaging will be performed using Visioscan® VC 20plus to take an image of the target lesion. The Visioscan software will be used to calculate the analyze the images for skin roughness (SEr, an increase in values indicates an improvement in roughness) and smoothness (SEsm, a decrease in values indicates an improvement in skin smoothness).
Subject treatment satisfaction | Week 2, Week 4, Week 8
  Subjects will be asked about their perception, satisfaction, and preference with each study treatment using a self-assessment questionnaire. Questionnaires will be tabulated; and the frequency and percentage of all response options will be reported for each question and time point. Favorable responses (i.e., strongly agree and agree, yes), neutral responses (i.e., neither agree nor disagree, no difference), and unfavorable responses (i.e., strongly disagree and disagree, no) will be tabulated and reported as appropriate. Percentage of favorable and unfavorable responses will be provided for each question.
Incidence of psoratic irritation [tolerability assessment] | Baseline, Week 2, Week 4, Week 8
  Tolerability assessment will be performed by the Investigator (parameter: dryness) and by subjects (parameters: burning/stinging and itching) using a 4-point analog scale (with half-point scores used as necessary to better describe the clinical condition). Investigator and subjects will grade the degree of irritation of target lesion areas on a scale of 0 to 3, with 0 meaning parameter is not present, and 3 meaning parameter is severely present. A decrease in scores or lack of significant increase indicates tolerability/safety of the treatment products.

SECONDARY OUTCOMES:
Subject Quality of Life Satisfaction | Baseline, Week 8
  Subjects will be asked about their life quality by completing a Quality of Life questionnaire. Each response will be assigned a numerical score, and all scores will be summed to determine the Dermatology Quality of Life Index. A decrease in score totals from baseline to Week 8 indicates an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, MD, Principal Investigator — Dermatology Consulting Services, High Point NC; George F Hougeir, MD, Principal Investigator — Southeast Dermatology Specialist, LLC
Locations (3):
- United States (3):
  - Southeast Dermatology Specialists, LLC, Columbus, Georgia
  - Southeast Dermatology Specialists, LLC, Douglasville, Georgia
  - Dermatology Consulting Services, High Point, North Carolina

IPD SHARING:
Plan to Share IPD: No